CLINICAL TRIAL: NCT02527226
Title: Post-parotidectomy Facial Paresis: Intraoperative and Postoperative Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eric J. Moore, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-004441
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Parotid Neoplasms; Facial Paralysis
MeSH Terms: conditions — Parotid Neoplasms; Facial Paralysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No facial exercises (No Intervention): This group will not receive any training in facial exercises.
- Facial exercises (Experimental): This group will receive instruction to perform a series of self-administered exercises of facial expression and movements.
  Interventions: Behavioral: Facial exercises

INTERVENTIONS:
Behavioral: Facial exercises — A series of self-administered facial movements and expressions.
  Arms: Facial exercises

SUMMARY:
This is a protocol to govern the prospective trial of facial nerve monitoring in patients undergoing parotidectomy with an eye towards interpreting if the facial nerve monitor provides useful information to operating surgeons and if the information provided by the facial nerve monitor can predict degrees of postoperative facial nerve paresis.

Additionally, the study will determine if performing daily facial rehabilitation exercises provides a benefit in reducing time to recovery of temporary post-parotidectomy paresis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Planned parotid gland surgery (superficial or total parotidectomy)
* Benign or malignant disease

Exclusion Criteria:

* Pregnancy
* Preoperative facial nerve dysfunction
* Revision operation
* History of preoperative radiation to the surgical field
* Entire nerve not dissected
* Intentional nerve sacrifice
* Poor signal to noise ratio during surgery
* Lack of access to device compatible with video conferencing software, or lack of access to broadband internet connection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Postoperative facial weakness | postoperative day 1
  Measure degree of facial weakness on postop day 1

SECONDARY OUTCOMES:
Time to resolution of facial weakness | 3 months
  Monitor time to resolution of weakness in the facial exercises and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Eric Moore, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota